CLINICAL TRIAL: NCT04391933
Title: MRI Staging in Colon Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MR Colon
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2020-05

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Sensitivity, specificity, positivity predictive values and negative predictive values are calculated form the histopathological surgical specimen. This will be the endpoint for both CT and MRI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI colon cancer (Other): MRI scan of patients with colon cancer
  Interventions: Diagnostic Test: MRI 3 tesla

INTERVENTIONS:
Diagnostic Test: MRI 3 tesla — MRI of colon cancer. Sensitivity, specificity, positivity predictive values and negative predictive values are calculated form the histopathological surgical specimen. This will be the endpoint for both CT and MRI.

SUMMARY:
The main purpose of this study is to investigate whether magnetic ressonance imaging (MRI) can be used in treatment planning with assessment of diagnostic accuracy. With the inclusion of 150 patients the study will investigate whether MRI is useful and better than CT scanning in patients with colon tumors. And also if MRI is useful after neoadjuvant treatment.

DETAILED DESCRIPTION:
Colon cancer is a frequent disease in Denmark with over 3200 new cases and about 1350 deaths per year.

CT scanning is currently the national standard method for determining the stage of disease planning for treatment. CT scan can sufficiently distinct between minor and advanced colon tumors. Prevalence of advanced tumors was well over 40% in the CT study from Vejle Hospital in 2013. Sensitivity and specificity of detection of advanced colon tumors in the CT study was approx. 70% and 80%, respectively. A small MRI pilot study showed higher sensitivity and specificity of 89% and 96%, respectively.

MRI scan is currently performed in most patients with rectal cancer, which has resulted in better treatment planning and increased survival. MRI scan of the rectum is documented with higher accuracy than CT scan. There has been reluctance to introduce MRI scan in patients with colon cancer, as the colon has more peristalsis than the rectum, and movement of the bowel can result in image quality reduction in MRI. However, in recent years MRI has become faster and thereby less sensitive to movements.

MRI scanning may in the future help to select the patients who will benefit from neoadjuvant treatment. In addition, with MRI it is possible to perform MRI diffusion measurements of the tumor, which gives an estimate of the tumor's cell density. It will also be possible to investigate whether this changes the MRI diffusion restriction during the neoadjuvant treatment.

This study is prospective and uses state of the art equipment with a 3 tesla MRI unit.

The main purpose of the study is to investigate whether MRI can be used in treatment planning with assessment of diagnostic accuracy. With the inclusion of 150 patients the study investigates whether MRI is useful and better than CT in patients with colon tumors. And also if MRI is useful after neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with colon cancer
* 18 years old or older
* Written and verbally informed consent

Exclusion Criteria:

* Pacemakers, implanted medical pumps, and nerve stimulators
* Cochlea implants and cerebral aneurism clips will in some cases be absolute contraindications to MRI examinations.
* Previous treatment with radiation and or chemotherapy
* Serious disease that contraindicates surgical treatment, including severe heart disease
* Any type of cancer other than of the colon (excluding skin cancer, cancer in situ, endometrial cancer, malignant melanoma)
* Any other condition or disease that from the investigator's point of view makes it inappropriate for the patient to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Is MRI usefull in colon cancer patients | 2 years
  Investigate the degree of accuracy in tumor stage compared to the histopathological surgical composition.

CONTACTS AND LOCATIONS:
Overall Officials: Søren R Rafaelsen, MD, DMSc, Study Chair — Vejle Hospital
Locations (1):
- Vejle Hospital, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: hospital — http://www.sygehuslillebaelt.dk/wm223295
- Available data/document: Informed Consent Form: CPR — https://komite.regionsyddanmark.dk/wm258128